CLINICAL TRIAL: NCT01269359
Title: Robotic Assisted Vertebral Body Augmentation - a Radiation Reduction Tool
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Yair Barzilay, Hadassah Medical Organization
Other Study IDs: BARZ-003HMO-CTIL
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Vertebral Body Augmentation
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- radiation
  Interventions: Procedure: robotic assisted surgery

INTERVENTIONS:
Procedure: robotic assisted surgery — Robotic guidance: SpineAssist™ (Mazor Surgical Technologies, Caesarea, Israel), is a bone-mounted miniature robot. It is a semi-active system offering surgical tool guidance while leaving performance of the actual surgical operation, such as the drilling, in the surgeon's hands.

SUMMARY:
Modern orthopedic and spine surgeons strive towards minimizing surgical exposure and towards increased precision in the placement of implants. This trend requires an increased use of fluoroscopic guidance, which leads to increased exposure of the patient, surgeon and the operating room staff to radiation.

Robotic assisted spine surgery is routinely performed in the authors' institution for a variety of indications such as degenerative conditions, trauma, tumors , infections and deformity correction11. The objective of this study is to compare the radiation exposure time during robotic guided vertebral body augmentation to the published results for similar surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Ages 18-85

Exclusion Criteria:

* Unwillingness to participate the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men and women that are candidates to vertebral body augmentation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
amount of radiation
  amount of radiation is calculated from the DLP (Dose Length Product)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organizaton, Jerusalem, Israel